CLINICAL TRIAL: NCT04746937
Title: Clinical Study to Evaluate the Possible Efficacy and Safety of Nitazoxanide in Secondary Prevention of Spontaneous Bacterial Peritonitis in Cirrhotic Patients
Brief Title: Nitazoxanide in Prevention of Secondary Spontaneous Peritonitis
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Eslam Mostafa Elasawy AlTaras, Clinical Pharmacist, Tanta University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: NTZ in Prevention of SBP
Record Dates: First submitted 2021-02-05; First posted 2021-02-10 (Actual); Last update posted 2021-02-10 (Actual); Status verified 2021-02

CONDITIONS: Spontaneous Bacterial Peritonitis
MeSH Terms: interventions — nitazoxanide; Norfloxacin

STUDY DESIGN:
Intervention Model Description: Randomized Double-Blind Placebo-Controlled study
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (Placebo Comparator): They will receive standard therapy plus placebo
  Interventions: Drug: Norfloxacin
- Nitazoxanide Group (Active Comparator): They will receive standard therapy plus nitazoxanide
  Interventions: Drug: Nitazoxanide; Drug: Norfloxacin

INTERVENTIONS:
Drug: Nitazoxanide — nitazoxanide adjuvant to standard therapy
  Other Names: NTZ
  Arms: Nitazoxanide Group
Drug: Norfloxacin — Standard therapy

SUMMARY:
the study is to evaluate the possible efficacy and safety of nitazoxanide as an adjuvant therapy in the secondary prevention of SBP in patient with cirrhosis.

DETAILED DESCRIPTION:
due to high recurrence rate of spontaneous bacterial peritonitis , we will study and evaluate the possible efficacy and safety of NTZ as an adjuvant therapy in the secondary prevention of SBP in patient with cirrhosis.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 21 - 65 years old with cirrhosis and ascites who had at least one previous confirmed episode of spontaneous bacterial peritonitis.

Exclusion Criteria:

* Exclusion criteria included active gastrointestinal bleeding Hepatic encephalopathy (>grade 2) Hepatocellular carcinoma (HCC) or other malignancies Allergy to used medications.

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-03 (Estimated); Primary Completion 2022-03 (Estimated); Study Completion 2022-05 (Estimated)

PRIMARY OUTCOMES:
Prevention of Secondary Spontaneous Bacterial Peritonitis | 3 months
  Reduction in incidence of secondary Spontaneous Bacterial Peritonitis (SBP) compared to control group

SECONDARY OUTCOMES:
Change in Biological Biomarkers | 3 months
  Measurement of Tumor necrosis factor alfa , Procalcitonin(PCT), C-Reactive protein(CRP) and Erythrocyte sedimentation rate(ESR) with further calculation of PEC index [PEC index = PCT × (ESR + CRP)] before and after trial period

CONTACTS AND LOCATIONS:
Overall Officials: Sahar M. Elhagar, Professor, Study Director — Supervisor for my master degree